CLINICAL TRIAL: NCT06680999
Title: Title Endovascular Treatment of Superior Cave Syndromes Reaching the Trifurcation: a Single-Center Case Series
Acronym: TESC-Tri
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0299
Record Dates: First submitted 2024-03-21; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Superior Cave Syndrome
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treated patients: All patients treated by endovascular surgery (stenting) at Hospices Civils de Lyon between March 2019 and July 2023 for superior cave syndrome, with lesions reaching the trifurcation (elective involvement of the superior vena cava)
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Preoperative, intraoperative and follow-up data collection: consultation and anesthesia reports, hospitalization reports and imaging data to evaluate the feasibility and efficacy of endovascular treatment of superior vena cava syndromes involving the trifurcation. Data collection will last 1 month and will be performed by a Vascular Surgery resident of the hospital.

SUMMARY:
Superior vena cava syndrome (SCS) is caused by obstruction of blood flow in the superior vena cava, which allows venous return from the upper half of the body to the heart.

The causes are most often oncological, but can also be benign (coagulopathy, Behçet) or iatrogenic (catheterisation, PAC).

The surgical management of superior vena cava syndromes (SCS) involves the use of innovative endovascular techniques, which have become the therapy of first choice for symptomatic patients, whether the occlusion occurs in a benign or malignant context. For occlusive lesions involving the trifurcation, there are several surgical approaches and strategies, but very little data on their efficacy. In particular, Y-stenting has been described in several case reports as a means of treating the SCS and keeping the two jugulo-subclavian veins (VJSC) patent. This innovative technique has been used for several years by the vascular surgery team at Hôpital Louis Pradel.

The aim of our study is to assess the feasibility and medium-term efficacy of innovative endovascular treatments for SCS involving the trifurcation.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated by endovascular surgery (stenting) at Hospices Civils de Lyon between March 2019 and July 2023 for superior cave syndrome

Exclusion Criteria:

* Minor patients
* Patients unable to give consent
* Patients unable to understand French
* Patients with lesions not reaching the trifurcation (elective involvement of the superior vena cava)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated by endovascular surgery (stenting) at Hospices Civils de Lyon between March 2019 and July 2023 for superior cave syndrome with lesions reaching the trifucation (elective involvement of the superior vena cava)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Technical success, immediate clinical success | The primary endpoint will be evaluated by : - Technical success defined by patency postoperatively and at 1 month follow-up confirmed by phleboscanner. Assessment of patency after revascularisation will be based on CT scan data (if possible) or on the r
  The primary endpoint will be evaluated by :
  - Technical success defined by patency postoperatively and at 1 month follow-up confirmed by phleboscanner.
  Assessment of patency after revascularisation will be based on CT scan data (if possible) or on the results of ultrasound data (letter from the angiologist) if this is the only test performed. Re-thrombosis of the inferior vena cava (IVC) or one of the two subclavian jugular veins (SCJV) will be sufficient to establish the absence of patency in our study.
  * Immediate clinical success defined by an improvement in symptoms observed by the medical team, and by a Yu score of less than or equal to 1 postoperatively and at 1 month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular and Endovascular Surgery Department, Hôpital Louis Pradel, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No